CLINICAL TRIAL: NCT02019082
Title: The Effect of Low-intensity Direct Current on the Expression of Vascular Endothelial Growth Factor and Nitric Oxide in Diabetic Foot Ulcers
Brief Title: Electrical Stimulation and Expression of VEGF and NO in Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: giti torkaman (Other)
Responsible Party: Sponsor-Investigator, giti torkaman, professor, Tarbiat Modarres University
Organization: Tarbiat Modarres University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: د 50/259
Record Dates: First submitted 2013-10-09; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrical stimulation (Active Comparator): electrical stimulation group, group who received direct current ES at sensory threshold intensity for 1 h/day, 3 days/week, for 4 weeks (12 sessions)
  Interventions: Device: Electrical Stimulation (BTL-5000 series, United Kingdom)
- placebo (Placebo Comparator): In the placebo group, the treatment procedure was the same as that the ES group, but the current intensity was zero.
  Interventions: Device: placebo

INTERVENTIONS:
Device: Electrical Stimulation (BTL-5000 series, United Kingdom) — Direct current ES
  Arms: electrical stimulation
Device: placebo — the intervention procedure was the same as that the ES group, but the current intensity was zero
  Arms: placebo

SUMMARY:
This study aimed to investigate the effect of low intensity cathodal direct current on the release of plasma vascular endothelial growth factor (VEGF) and nitric oxide (NO) in diabetic foot ulceration.

DETAILED DESCRIPTION:
Twenty type 2 diabetic patients with foot ulceration and 13 age-matched healthy subjects were enrolled. Patients were randomly assigned to electrical stimulation (ES, n=10) or sham ES (placebo, n=10) groups. ES group received cathodal direct current for 1 h/day, 3 days/week, for 4 weeks (12 sessions). Blood sample was collected for VEGF and NO measurement in the first and last treatment sessions before and after intervention. Wound surface area (WSA) and skin temperature were measured at 1st, 6th, and 12th session.

ELIGIBILITY:
Inclusion Criteria:

* Wagner classification DFU 2;
* age 40-60 years;
* mild to moderate diabetic neuropathy;
* ABI>0.7
* wound surface area>1.5cm2

Exclusion Criteria:

* fracture in a lower limb,
* a severe infection,
* a malignancy,
* kidney failure,
* skin diseases,
* osteomyelitis,
* pregnancy,

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The plasma level of VEGF(pg/ml) and NO (microM) | prior to the 1st electrical stimulation session(day 1) and 1 hour later, and prior to the 12th electrical stimulation session(day 26) and 1 hour later

SECONDARY OUTCOMES:
skin temperature (degree of centigrade) | prior the 1st electrical stimulation session (day 1) and 1 hour later
skin temperature (degree of centigrade) | prior the 6th electrical stimulation session (day 12) and 1 hour later
skin temperature (degree of centigrade) | prior the 12th electrical stimulation session (day 26) and 1 hour later
Wound surface area(cm2) | on day 1, 12, and 26

CONTACTS AND LOCATIONS:
Overall Officials: giti torkaman, PhD, Study Director — professor of physical therapy, physical therapy department, faculty of medical sciences, tarbiat modares univercity
Locations (1):
- Physical Therapy Department, Faculty of Medical Sciences, Tehran, Iran